CLINICAL TRIAL: NCT00754572
Title: A Single-arm, Open-label Study of the Safety and Reduction of Signs and Symptoms During Treatment With Tocilizumab in Combination With Methotrexate, in Patients With Moderate to Severe Active Rheumatoid Arthritis
Brief Title: A Study to Assess the Effect of Tocilizumab Plus Methotrexate on Safety and Signs and Symptoms in Patients With Moderate to Severe Active Rheumatoid Arthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML21530
Record Dates: First submitted 2008-09-17; First posted 2008-09-18 (Estimated); Results first posted 2015-05-15 (Estimated); Last update posted 2015-05-15 (Estimated); Status verified 2015-05

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — tocilizumab; Methotrexate

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: tocilizumab [RoActemra/Actemra]; Drug: methotrexate

INTERVENTIONS:
Drug: tocilizumab [RoActemra/Actemra] — 8mg/kg iv, every 4 weeks
Drug: methotrexate — 10-25mg oral or parenteral weekly.

SUMMARY:
This single arm, open-label study will assess the safety and efficacy with regar d to reduction of signs and symptoms of treatment with tocilizumab in combinatio n with methotrexate, in patients with moderate to severe active rheumatoid arthr itis. Patients will receive tocilizumab 8mg/kg iv, every 4 weeks and methotrexat e 10-25mg weekly. The anticipated time on study treatment is 3-12 months, and th e target sample size is <500 individuals.

ELIGIBILITY:
Inclusion Criteria:

* patients >=18 years with moderate to severe active RA for at least 6 months;
* swollen joint count >=6 (66 joint count) and tender joint count >=8 (68 joint count) at screening;
* inadequate response to stable dose of MTX;
* patients of reproductive potential must be using a reliable means of contraception.

Exclusion Criteria:

* rheumatic autoimmune disease other than RA;
* patients with functional class IV RA;
* diagnosis of juvenile idiopathic or rheumatoid arthritis before age 16 or a history of current inflammatory joint disease other than RA;
* prior treatment failure with anti-tumor necrosis factor agent;
* pregnant or breastfeeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 418 (Actual)
Dates: Start 2009-02; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (51):
- Argentina (4):
  - Buenos Aires
  - Córdoba
  - San Miguel
  - San Miguel de Tucumán
- Brazil (18):
  - Fortaleza, Ceará
  - Vitória, Espírito Santo
  - Salvador, Estado de Bahia
  - Brasília, Federal District
  - Belo Horizonte, Minas Gerais
  - Juiz de Fora, Minas Gerais
  - Curtiba, Paraná
  - Recife, Pernambuco
  - Rio de Janeiro, Rio de Janeiro
  - Caxias do Sul, Rio Grande do Sul
  - Porto Alegre, Rio Grande do Sul
  - Florianópolis, Santa Catarina
  - Botucatu, São Paulo
  - Campinas, São Paulo
  - Ribeirão Preto, São Paulo
  - Santo André, São Paulo
  - São José do Rio Preto, São Paulo
  - São Paulo, São Paulo
- Chile (3):
  - Concepción
  - Santiago
  - Temuco
- Colombia (6):
  - Barranquilla
  - Bogotá
  - Bucaramanga
  - Cali
  - Chia-Cundinamarca
  - Medellín
- Costa Rica (3):
  - Cartago
  - Heredia
  - San José
- Ecuador (3):
  - Cuenca
  - Guayaquil
  - Quito
- Mexico (6):
  - Chihuahua City
  - Guadalajara
  - Mexico City
  - Miexico City
  - Querétaro
  - San Luis Potosí City
- Peru (4):
  - Arequipa
  - Jesus Maria
  - Lima
  - San Isidro
- Montevideo, Uruguay
- Venezuela (3):
  - Barquisimeto
  - Caracas
  - Maracaibo

RESULTS

PARTICIPANT FLOW:
Groups:
- Tocilizumab: Participants received tocilizumab 8 milligrams per kilogram (mg/kg) intravenously (iv), once every 4 weeks for a total of 6 infusions along with methotrexate 10-25 mg weekly, orally or parenterally. The dose of methotrexate should have remained stable throuhgout the study.
Period: Overall Study
Arm/Group | Tocilizumab
Started | 418
Completed | 347
Not Completed | 71
Not completed — Adverse Event | 19
Not completed — Other | 39
Not completed — Protocol Violation | 3
Not completed — Withdrawal by Subject | 3
Not completed — Lack of Efficacy | 2
Not completed — Death | 1
Not completed — Administrative Reason | 3
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Population: Intention to treat (ITT) population: All participants who received at least one dose of study drug and who had at least one effectiveness measurement performed after baseline.
Groups:
- Tocilizumab: Participants received tocilizumab 8 mg/kg iv, once every 4 weeks for a total of 6 infusions along with methotrexate 10-25 mg weekly, orally or parenterally. The dose of methotrexate should have remained stable throughout the study.
Arm/Group | Tocilizumab
Number analyzed (Participants) | 418
Age, Continuous [Mean (Standard Deviation); unit: years] | 48.69 (12.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 371
  Male | 47

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With American College of Rheumatology (ACR) 50 Response at Week 24
Description: ACR50 is defined as 50 percent (%) improvement in: a) Swollen Joints Count (SJC) and Tender Joints Count (TJC) and b) Three of the following 5 assessments:
  1. Participant's global assessment of pain by Visual Analog Scale (VAS)
  2. Participant's global assessment of disease activity (VAS)
  3. Investigator/Physician's global assessment of disease activity (VAS)
  4. Participant's assessment of disability measured by the Health Assessment Questionnaire Disability Index (HAQ-DI)
  5. Acute phase reactant levels - Erythrocyte Sedimentation Rate or C-Reactive Protein (ESR or CRP)
Time Frame: Week 24
Population: ITT Population; All participants with endpoint values collected at Week 24 were included in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 381
percentage of participants | 73.23 [68.78 to 77.67]

2. Secondary Outcome: Percentage of Participants With ACR20 and ACR70 Response at Week 24
Description: ACR20 and ACR70 are defined as 20 and 70 percent improvement respectively in: a) SJC and TJC and b) Three of the following 5 assessments:
  1. Participant's global assessment of pain by VAS
  2. Participant's global assessment of disease activity (VAS)
  3. Investigator/Physician's global assessment of disease activity (VAS)
  4. Participant's assessment of disability measured by HAQ-DI
  5. Acute phase reactant (ESR or CRP)
Time Frame: Week 24
Population: ITT Population; All participants with endpoint values collected at Week 24 were included in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 381
percentage of participants
  ACR 20 | 90.55 [87.61 to 93.49]
  ACR 70 | 50.39 [45.37 to 55.41]

3. Secondary Outcome: Time to Onset of ACR20, ACR50, and ACR70
Description: ACR20, ACR50 and ACR70 are defined as 20, 50 and 70 percent improvement respectively in: a) SJC and TJC and b) Three of the following 5 assessments:
  1. Participant's global assessment of pain by VAS
  2. Participant's global assessment of disease activity (VAS)
  3. Investigator/Physician's global assessment of disease activity (VAS)
  4. Participant's assessment of disability measured by HAQ-DI
  5. Acute phase reactant (ESR or CRP)
Time Frame: Baseline and Week 24
Population: Data were not analyzed because of inconsistencies in the pooled data between countries.
Arm/Group | Tocilizumab
Number analyzed (Participants) | 0

4. Secondary Outcome: Change From Baseline in Hemoglobin at Week 24
Time Frame: Baseline and Week 24
Population: Data were not analyzed because of inconsistencies in the pooled data between countries.
Arm/Group | Tocilizumab
Number analyzed (Participants) | 0

5. Secondary Outcome: SJC and TJC at Baseline and Week 24
Description: The number of swollen joints (66 joint count) were scored as swollen=1 and not swollen=0, and the number of tender joints (68 joint count ) were scored as tender=1 and not tender=0, and counted. Scores ranged from 0 to 66 for swollen joint counts and from 0 to 68 for tender joint counts. A positive change from baseline represents an improvement (a reduction in the number of swollen or tender joints).
Time Frame: Baseline and Week 24
Population: ITT Population; All participants with endpoint values collected at both baseline and Week 24 were included in the analysis.
Measure: Mean (Standard Deviation); unit: joints
Arm/Group | Tocilizumab
Number analyzed (Participants) | 384
joints
  TJC-Baseline | 25.06 (13.83)
  TJC-Week 24 | 4.57 (7.57)
  SJC-Baseline | 16.09 (8.69)
  SJC-Week 24 | 2.56 (4.26)

6. Secondary Outcome: Percent Change From Baseline in SJC and TJC at Week 24
Description: as for outcome 5
Time Frame: Baseline and Week 24
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Tocilizumab
Number analyzed (Participants) | 384
percent change
  TJC | 81.2 (28.1)
  SJC | 84.8 (22.5)

7. Secondary Outcome: Pain as Assessed by the Participant at Baseline and Week 24
Description: The participants assessed their pain using a 0 to 100 millimeter (mm) VAS. The left-hand extreme of the line equals 0 mm, and is described as "no pain" and the right-hand extreme equals 100 mm as "unbearable pain". The participants marked the line corresponding to the level of their pain and the distance from the left edge was measured. A positive change from baseline represents an improvement.
Time Frame: Baseline and Week 24
Population: ITT Population; All participants with endpoint values collected at the specified timepoints were included in the analysis. number (n) equals (=) number of participants analyzed for the given parameter at the specified time point.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Tocilizumab
Number analyzed (Participants) | 384
mm
  Baseline (n=384) | 68.01 (20.39)
  Week 24 (n=381) | 22.94 (22.53)

8. Secondary Outcome: Percent Change From Baseline in Pain as Assessed by the Participant at Week 24
Description: as for outcome 7
Time Frame: Baseline and Week 24
Population: ITT Population; All participants with endpoint values collected at Baseline and Week 24 were included in the analysis.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Tocilizumab
Number analyzed (Participants) | 381
percent change | 54.2 (177.0)

9. Secondary Outcome: Participant's Global Assessment of Disease Activity at Baseline and Week 24
Description: The participant's global assessment of disease activity is assessed on a 0 to 100 mm horizontal VAS by the participant. The left-hand extreme of the line equals 0 mm, and is described as "no disease activity" (symptom-free and no arthritis symptoms) and the right-hand extreme equals 100 mm, as "maximum disease activity" (maximum arthritis disease activity). A positive change from baseline represents an improvement (reduced level of disease activity).
Time Frame: Baseline and Week 24
Population: ITT Population. All participants with endpoint values collected at the specified timepoints were included in the analysis. n= number of participants analyzed for the given parameter at the specified time point.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Tocilizumab
Number analyzed (Participants) | 384
mm
  Baseline (n=384) | 69.46 (20.84)
  Week 24 (n=381) | 23.60 (22.68)

10. Secondary Outcome: Percent Change From Baseline in Participant's Global Assessment of Disease Activity at Week 24
Description: as for outcome 9
Time Frame: Baseline and Week 24
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Tocilizumab
Number analyzed (Participants) | 381
percent change | 61.7 (43.1)

11. Secondary Outcome: Physician's Global Assessment of Disease Activity at Baseline and Week 24
Description: The physician's global assessment of disease activity is assessed on a 0 to 100 mm VAS by the physician. The left-hand extreme of the line equals 0 mm, and is described as "no disease activity" (symptom-free and no arthritis symptoms) and the right-hand extreme equals 100 mm as "maximum disease activity" (maximum arthritis disease activity). The physicians marked the line corresponding to their assessment and the distance from the left edge was measured. A positive change from baseline represents an improvement (reduced level of disease activity).
Time Frame: Baseline and Week 24
Population: ITT Population. All participants with endpoint values collected at the specified timepoints were included in the analysis. n=number of participants analyzed for the given parameter at the specified visit.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Tocilizumab
Number analyzed (Participants) | 384
mm
  Baseline (n=384) | 67.32 (16.64)
  Week 24 (n=381) | 17.92 (18.16)

12. Secondary Outcome: Percent Change From Baseline in Physician's Global Assessment of Disease Activity at Week 24
Description: as for outcome 11
Time Frame: Baseline and Week 24
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Tocilizumab
Number analyzed (Participants) | 381
percent change | 71.2 (38.7)

13. Secondary Outcome: HAQ-DI at Baseline and Week 24
Description: HAQ-DI includes 20 questions concerning participant's activities of daily life, grouped in 8 scales of 2 to 3 questions for each activity. To respond to each question, a four-level response (score of 0 to 3 points), with higher scores showing larger functional limitations, was chosen. Scoring was as follows with respect to performance of participant's everyday activities: 0 =without difficulties; 1= with some difficulties; 2=with great difficulties; and 3= unable to perform these actions at all. Minimum score was 0, maximum score was 3. A positive change from baseline represents an improvement (reduced level of impairment).
Time Frame: Baseline and Week 24
Population: ITT Population. All participants with endpoint values collected at the specified timepoints were included in the analysis. n=number of participants analyzed for the given parameter at the specified time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 384
units on a scale
  Baseline (n=384) | 1.70 (0.63)
  Week 24 (n=376) | 0.79 (0.68)

14. Secondary Outcome: Percent Change From Baseline in HAQ-DI at Week 24
Description: HAQ-DI includes 20 questions concerning participant's activities of daily life, grouped in 8 scales of 2 to 3 questions for each activity. To respond to each question, a four-level response (score of 0 to 3 points), with higher scores showing larger functional limitations, was chosen. Scoring was as follows with respect to performance of participant's everyday activities: 0=without difficulties; 1=with some difficulties; 2=with great difficulties; and 3=unable to perform these actions at all. Minimum score was 0, maximum score was 3. A positive change from baseline represents an improvement (reduced level of impairment).
Time Frame: Baseline and Week 24
Population: ITT Population. All participants with endpoint values collected at both baseline and Week 24 were included in the analysis.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Tocilizumab
Number analyzed (Participants) | 376
percent change | 52.0 (49.3)

15. Secondary Outcome: Area Under The Curve (AUC) of the ACR(n)
Description: ACR-n was defined as the lowest of 3 values (the percent change in the swollen joint count, the percent change in the tender joint count, and the median of the other 5 measures in the ACR core data set which included Participant's global assessment of pain (VAS), Participant's global assessment of disease activity (VAS), Investigator/Physician's global assessment of disease activity (VAS), Participant's assessment of disability measured by the HAQ-DI Acute phase reactant levels - ESR or CRP). Therefore, a percentage value was assigned to each participant at each timepoint. AUC was calculated for each participant from baseline to Week 112. Mean and standard deviation values are are provided in percent*years.
Time Frame: Baseline and Weeks 2, 4, 8, 12, 16, 20 and 24
Population: ITT Population; All participants with endpoint values collected were included in the analysis.
Measure: Mean (Standard Deviation); unit: percent*years
Arm/Group | Tocilizumab
Number analyzed (Participants) | 391
percent*years | 20.8 (9.4)

16. Secondary Outcome: Percentage of Participants Achieving ACR20 Response
Description: ACR20 is defined as 20% improvement in: a) SJC and TJC and b) Three of the following 5 assessments:
  1. Participant's global assessment of pain (VAS)
  2. Participant's global assessment of disease activity (VAS)
  3. Investigator/Physician's global assessment of disease activity (VAS)
  4. Participant's assessment of disability measured by the HAQ-DI
  5. Acute phase reactant levels - ESR or CRP
Time Frame: Week 2
Population: ITT Population; All participants with endpoint values collected at Week 2 were included in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 389
percentage of participants | 40.10 [35.23 to 44.97]

17. Secondary Outcome: Odds Estimates for ACR Positive Response in Generalized Estimating Equation (GEE) Models
Description: The probability of ACR positive response was determined using the GEE.
Time Frame: Weeks 2, 4, 8, 12, 16, 20, 24
Population: ITT Population; All participants with endpoint values collected were included in the analysis.
Measure: Number (95% Confidence Interval); unit: odds
Arm/Group | Tocilizumab
Number analyzed (Participants) | 418
odds
  Week 2 Odds ACR50 | 0.10 [0.07 to 0.14]
  Week 4 Odds ACR50 | 0.33 [0.27 to 0.42]
  Week 8 Odds ACR50 | 0.87 [0.72 to 1.05]
  Week 12 Odds ACR50 | 1.39 [1.14 to 1.69]
  Week 16 Odds ACR50 | 1.55 [1.28 to 1.89]
  Week 20 Odds ACR50 | 1.86 [1.52 to 2.27]
  Week 24 Odds ACR50 | 2.39 [1.93 to 2.95]
  Week 2 Odds ACR20 | 0.63 [0.51 to 0.76]
  Week 4 Odds ACR20 | 1.50 [1.24 to 1.83]
  Week 8 Odds ACR20 | 4.80 [3.73 to 6.19]
  Week 12 Odds ACR20 | 4.80 [3.73 to 6.19]
  Week 16 Odds ACR20 | 4.65 [3.61 to 5.97]
  Week 20 Odds ACR20 | 6.46 [4.88 to 8.56]
  Week 24 Odds ACR20 | 6.88 [5.16 to 9.18]
  Week 4 Odds ACR70 | 0.08 [0.06 to 0.12]
  Week 8 Odds ACR70 | 0.27 [0.21 to 0.34]
  Week 12 Odds ACR70 | 0.41 [0.34 to 0.51]
  Week 16 Odds ACR70 | 0.53 [0.44 to 0.65]
  Week 20 Odds ACR70 | 0.75 [0.62 to 0.91]
  Week 24 Odds ACR70 | 0.92 [0.76 to 1.12]

18. Secondary Outcome: Change From Baseline in Disease Activity Score Based on 28 Joint Count (DAS28) at Week 24
Description: DAS28 calculated from the number of SJC and TJC using the 28 joints count, the ESR (mm/hour) and participant's global assessment of disease activity (participant rated arthritis activity assessment with transformed scores ranging 0 to 10; higher scores indicated greater affectation due to disease activity). DAS28 (less than or equal to ) ≤3.2 = low disease activity, DAS28 (greater than) >3.2 to 5.1 = moderate to high disease activity.
Time Frame: Baseline and Week 24
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 399
score on a scale | 4.4 (1.6)

19. Secondary Outcome: Percentage of Participants With a Response by Categorical DAS28 Responses According to The European League Against Rheumatism (EULAR Response) at Week 24
Description: DAS28- based EULAR response criteria were used to measure individual response as none, good, and moderate, depending on the extent of change from baseline and the level of disease activity reached. Good response: change from baseline >1.2 with DAS28 < 3.2; moderate response: change from baseline >1.2 with DAS28 >3.2 to <5.1 or change from baseline >0.6 to <1.2 with DAS28 <5.1; No response: change from baseline < 0.6 or change from baseline >0.6 and <1.2 with DAS28 >5.1.
Time Frame: Week 24
Population: ITT Population; All participants with endpoint values collected at Week 24 were included in the analysis.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 399
Percentage of Participants
  Good Response | 68.17 [63.60 to 72.74]
  Moderate Response | 29.57 [25.10 to 34.05]
  No Response | 2.26 [0.80 to 3.71]

20. Secondary Outcome: AUC of DAS28
Description: The AUC was computed using the trapezoidal rule, considering baseline value as 0, through NCSS software. For each participant, AUC for DAS28 units was calculated. Each individual AUC DAS28 value was divided by 52 to have the conversion of AUC DAS28 in unit weeks to AUC DAS28 in unit years, as 1 week is approximately 1/52 years. The set of individual AUC DAS28 was computed as summary statistics.
Time Frame: Weeks 2, 4, 8, 12, 16, 20 and 24
Population: ITT Population; All participants with endpoint values collected were included in the analysis.
Measure: Mean (Standard Deviation); unit: scores on a scale * years
Arm/Group | Tocilizumab
Number analyzed (Participants) | 416
scores on a scale * years | 11.8 (4.2)

21. Secondary Outcome: Fatigue as Assessed Using the Functional Assessment of Chronic Illness Therapy (FACIT-Fatigue) Score at Week 24
Description: FACIT-F is a 13-item questionnaire. Participants scored each item on a 5-point scale: 0 (Not at all) to 4 (Very much). The larger the participant's response to the questions (with the exception of 2 negatively stated), the greater the participant's fatigue. The sum of all responses resulted in the FACIT-Fatigue score for a total possible score of 0 (worse score) to 52 (better score). A higher score reflects an improvement in the participant's health status.
Time Frame: Week 24
Population: ITT Population. All participants with endpoint values collected at Week 24 were included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 403
score on a scale | 39.9 (9.4)

22. Secondary Outcome: Percentage of Participants Achieving Remission (DAS28 Less Than [<] 2.6) at Week 24
Description: DAS28 calculated from the SJC and TJC using the 28 joints count, the ESR (mm/hour) and participant's global assessment of disease activity (participant rated arthritis activity assessment with transformed scores ranging 0 to 10; higher scores indicated greater affectation due to disease activity). DAS28 (less than or equal to ) ≤3.2 = low disease activity, DAS28 (greater than) >3.2 to 5.1 = moderate to high disease activity and DAS28<2.6 = remission
Time Frame: Week 24
Population: ITT Population; All participants with endpoint values collected at Week 24 were included in the analysis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tocilizumab
Number analyzed (Participants) | 409
percentage of participants | 48.41 [43.57 to 53.25]

23. Secondary Outcome: Quality of Life (QoL) Assessed by Short-Form 36 (SF-36) at Week 24
Description: SF-36 is a standardized survey evaluating 8 aspects of functional health and well-being: physical and social functioning, physical and emotional role limitations, bodily pain, general health, vitality, and mental health. Total of 3 variables were analyzed (2 composite subscales and vitality score). The score for a section is an average of the individual question scores, which are scaled 0-100 (100=highest level of functioning).
Time Frame: Week 24
Population: ITT Population; All participants with endpoint values collected at Week 24 were included in the analysis.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tocilizumab
Number analyzed (Participants) | 378
score on a scale
  General Health | 42.5 (12.9)
  Physical functioning | 63.0 (24.2)
  Role limitations due to physical health | 64.0 (23.9)
  Role limitations due to emotional problems | 66.0 (24.1)
  Energy/fatigue | 48.9 (10.6)
  Emotional well-being | 54.5 (10.3)
  Social functioning | 38.2 (12.7)
  Pain | 63.6 (24.8)

24. Secondary Outcome: Mean Change in Rheumatoid Factor (RF) at Week 24 in Participants With Positive RF
Time Frame: Baseline and Week 24
Population: Data were not analyzed because of inconsistencies in the pooled data between countries.
Arm/Group | Tocilizumab
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse events were recorded from the date of first dose of drug administration until the end of study
Arm/Group | Tocilizumab
Serious Adverse Events (participants affected / at risk) | 30/418
Other Adverse Events (participants affected / at risk) | 324/418
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tocilizumab (N=418)
Pneumonia (Infections and infestations) | 3
Hypersensitivity (Immune system disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 1
Bradicardia (Cardiac disorders) | 1
Bronchitis (Infections and infestations) | 1
Chronic gastrointestinal bleeding (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Pyelonephritis acute NOS (Renal and urinary disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Septic shock (Infections and infestations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Headache (Nervous system disorders) | 1
Leukopenia NOS (Blood and lymphatic system disorders) | 2
Appendicitis (Infections and infestations) | 1
Asthmatic crisis (Respiratory, thoracic and mediastinal disorders) | 1
Herpes zoster (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 3
Urticaria (Skin and subcutaneous tissue disorders) | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1
Intervertebral disc herniation (Musculoskeletal and connective tissue disorders) | 1
Intervertebral discitis (Musculoskeletal and connective tissue disorders) | 1
Tendon rupture (Injury, poisoning and procedural complications) | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1
Fracture (Injury, poisoning and procedural complications) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Abscess (General disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tocilizumab (N=418)
Hypercholesterolemia (Metabolism and nutrition disorders) | 71
Hepatic enzyme increased (Investigations) | 70
Headache (Nervous system disorders) | 41
Urinary tract infection (Infections and infestations) | 41
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 39
Hypertension (Vascular disorders) | 32
Influenza (Infections and infestations) | 32
Pharyngitis (Infections and infestations) | 30
Leukopenia NOS (Blood and lymphatic system disorders) | 25
Back pain (Musculoskeletal and connective tissue disorders) | 22
Nausea (Gastrointestinal disorders) | 22
Stomatitis (Gastrointestinal disorders) | 22
Neutropenia (Blood and lymphatic system disorders) | 21
Blood bilirubin increased (Investigations) | 19
Upper respiratory tract infection (Infections and infestations) | 19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The study being conducted under this agreement is part of the overall study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the study, but after the first publication or presentation that involves the overall study. Sponsor may request that confidential information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.